CLINICAL TRIAL: NCT01308060
Title: A Multi-center Randomized, Double-blind, Placebo Controlled, Parallel-group Study of CD07743 for the Improvement of Lateral Canthal Lines (Crow's Feet)
Brief Title: A Multi-Center Study Of CD07743 for the Improvement of Lateral Canthal Lines (CROW'S FEET)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.03.SPR.40131
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2012-08

CONDITIONS: Canthal Lines
Keywords: Canthal lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin type A (Experimental): During part A, efficacy and safety parameters will be assessed for Azzalure vs. placebo
  Interventions: Drug: Botulinum Toxin Type A
- Placebo (Placebo Comparator): During part A, efficacy and safety parameters will be assessed for Azzalure vs. placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A — During part A, Azzalure will be administered at Baseline 60 Speywood units at canthal lines and compared with placebo.
  Arms: Botulinum Toxin type A
Other: Placebo
  Arms: Placebo

SUMMARY:
This double-blind study has two parts for each subject (same population):

Part A: initial treatment in Lateral Canthal Lines (LCL) (placebo-controlled):

* To assess the efficacy and safety of Azzalure® compared to placebo in the improvement of moderate to severe LCLs.
* To assess the subjects' level of satisfaction with the appearance of their LCLs compared to placebo.

Part B: repeated treatment in LCL with or without Glabellar Lines (GL) (active treatment, up to 1 year):

* To assess safety of Azzalure® following repeated administration in the improvement of moderate to severe LCLs.
* To assess the safety of Azzalure® when used concomitantly for improvement of moderate to severe LCLs and GLs.
* To assess the subjects' level of satisfaction with the appearance of their LCLs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 65 years of age (Screening visit),
* Moderate or severe (grade 2 or 3, Hund 2006) Lateral Canthal Lines "at maximum smile" determined by investigator at screening and baseline
* Mild to severe (grade 1, 2 or 3, Hund 2006) Lateral Canthal Lines "at rest" determined by investigator at screening and baseline
* The subject is a female of childbearing potential and has a negative urine pregnancy test (UPT) at screening and baseline
* Subjects who are not satisfied with their appearance at screening and baseline
* The subject is willing and able to comply with the requirements of the protocol and agree to adhere to the visit schedule, concomitant therapy prohibitions and must be compliant to the study instruction.
* The subject agrees to participate in the study, verified by dating and signing an approved written Informed Consent Form (ICF) and Photography Consent Form (PCF) (selected sites only if applicable) at the enrolment visit before any study procedures at screening

Exclusion Criteria:

* Any prior surgery affecting the orbicularis oculi muscle, prior blepharoplasty or brow lift, or any prior cosmetic procedures or scars that may interfere with the evaluation of the investigator.
* Previous insertion of any permanent, semi-permanent or biodegradable material in the periorbital region or facial treatment with augmentation material (e.g. silicon injections, collagen type implants, hyaluronic acid, lactic acid, etc.) within 12 months prior to screening.
* Any prior treatment with botulinum toxin (of any serotype)
* Previous treatment with lasers for skin resurfacing (e.g. CO2 (carbon dioxide)-laser) or treatment with deep chemical peels and any other esthetic or dermatologic treatments or procedures in any area of the face within 12 months prior to screening.
* Any planned facial cosmetic surgery or procedures during the study period.
* Presence of any bleeding disorders
* Pregnant or lactating women or women who are planning pregnancy during the study.
* Known hypersensitivity to any of the test materials or related compounds.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin Type A; Placebo: During part A, efficacy and safety parameters will be assessed for Azzalure vs. placebo
  Botulinum Toxin Type A: During part A, Azzalure will be administered at Baseline 60 Speywood units at canthal lines and compared with placebo.
  Part B was open-label, active treatment to all participants up to 1 year. (Therefore, "reason withdrawn" cannot be specified per group.)
Period: Part A
Arm/Group | Botulinum Toxin Type A | Placebo
Started | 252 | 83
Completed | 238 | 77
Not Completed | 14 | 6
Period: Part B
Arm/Group | Botulinum Toxin Type A | Placebo
Started | 238 | 77
Completed | 219 | 69
Not Completed | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Placebo: During part A, efficacy and safety parameters will be assessed for Azzalure vs. placebo
  Botulinum Toxin Type A: During part A, Azzalure will be administered at Baseline 60 Speywood units at canthal lines and compared with placebo.
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Placebo | Total
Number analyzed (Participants) | 252 | 83 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (8.6) | 49.3 (8.1) | 48.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 74 | 308
  Male | 18 | 9 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 249 | 83 | 332
  Hispanic | 1 | 0 | 1
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Germany | 121 | 39 | 160
  France | 92 | 31 | 123
  United Kingdom | 39 | 13 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders on the Severity of Lateral Canthal Lines "at Maximum Smile".
Description: A positive response (responder) is defined as a grade of 0 or 1 (none or mild), as assessed by the investigator.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 252 | 83
Participants | 119 | 6

2. Secondary Outcome: Number of Participants Satisfied With the Appearance of Their Lateral Canthal Lines
Description: Participants were asked to assess their degree of satisfaction with the appearance of their lateral canthal lines using a 4-point scale with the grades Very satisfied, Satisfied, Dissatisfied, and Very dissatisfied. A participant is considered satisfied if he/she answers Very satisfied or Satisfied.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 252 | 83
Participants | 165 | 14

ADVERSE EVENTS:
Description: Total Number at Risk in Arm "Botulinum Toxin Type A-Part B" is not consistent with the number in the Participant Flow for Part B since 11 subjects were ongoing in Part A at Day 85 when the Adverse Event (AE) summary for Part B begins; 326 were ongoing at Day 85 but only 315 received retreatment (which is when Part B started for an individual subject).
  AEs were collected together for Part B and recorded AEs cannot be attributed to specific interventions for this Part (all received active).
Groups:
- Botulinum Toxin Type A - Part A: During part A, efficacy and safety parameters will be assessed for Azzalure vs. placebo.
  Botulinum Toxin Type A: During part A, Azzalure will be administered at Baseline 60 Speywood units at canthal lines and compared with placebo.
- Placebo - Part A: During part A, efficacy and safety parameters will be assessed for Azzalure vs. placebo.
- Botulinum Toxin Type A - Part B: Part B was open-label, active treatment to all participants up to 1 year. The retreatment, or first treatment if randomized to placebo, injection defines for each subject the start of Part B.
Arm/Group | Botulinum Toxin Type A - Part A | Placebo - Part A | Botulinum Toxin Type A - Part B
All-Cause Mortality (participants affected / at risk) | 0/252 | 0/83 | 0/326
Serious Adverse Events (participants affected / at risk) | 5/252 | 1/83 | 11/326
Other Adverse Events (participants affected / at risk) | 0/252 | 0/83 | 0/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin Type A - Part A (N=252) | Placebo - Part A (N=83) | Botulinum Toxin Type A - Part B (N=326)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness transitory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes